CLINICAL TRIAL: NCT00419718
Title: Effect of Exercise on the Pharmacokinetics and Pharmacodynamics of Inhaled Human Insulin in Subjects With Type 1 Diabetes
Brief Title: Effect of Exercise on the Absorption of Inhaled Human Insulin in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1998-1562
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: inhaled human insulin

SUMMARY:
The trial is conducted in Europe. This clinical pharmacology trial investigates the effect of exercise on the pharmacokinetics and pharmacodynamics of inhaled insulin in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes more than or equal to 12 months
* Baseline HbA1c less than or equal to 11%
* Body mass index (BMI) less than or equal to 29 kg/m2
* Normal lung volumes
* Treatment with intensified insulin therapy for at least 3 months

Exclusion Criteria:

* Any present or history of pulmonary disease
* Any findings from the cardiopulmonary exercise test compromising safety of moderate exercise
* Impaired hepatic or renal function
* Cardiac problems
* Uncontrolled hypertension
* Current proliferative retinopathy or maculopathy
* Treatment with drugs, which may interfere with insulin action, glucose metabolism or recovery from hypoglycaemia (judged by investigator)
* Current smoking or smoking within the last 6 months
* Blood donation (more than 500 mL) within the last nine weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-10; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma insulin profile in the interval | From 30-150 min after trial product administration

SECONDARY OUTCOMES:
Area under the plasma insulin profile in the interval from 120-240 min after trial product administration
Area under the plasma insulin profile in the interval from 240-360 min after trial product administration
Area under the plasma insulin profile in the interval 0-600 min after trial product administration
Maximum plasma insulin concentration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

REFERENCES:
- [Result] Petersen AH, Kohler G, Korsatko S, Wutte A, Wonisch M, Jeppesen OK, Sparre T, Clauson P, Laursen T, Wollmer P, Pieber TR. The effect of exercise on the absorption of inhaled human insulin via the AERx insulin diabetes management system in people with type 1 diabetes. Diabetes Care. 2007 Oct;30(10):2571-6. doi: 10.2337/dc06-2589. Epub 2007 Jul 9. PMID 17620446
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com